CLINICAL TRIAL: NCT00671099
Title: Tachikawa Project for Prevention of Posttraumatic Stress Disorder With Polyunsaturated Fatty Acid (TPOP): TPOP-02 Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Japan Science and Technology Agency (Other)
Collaborators: University of Toyama (Other); Chiba University (Other)
Responsible Party: Principal Investigator, Yutaka Matsuoka, Psychiatrist, Japan Science and Technology Agency
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NDMC-TPOP-02
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Trauma; Posttraumatic Stress Disorder
Keywords: Patients; with high-energy; admitted; intensive care unit; motor vehicle accident; falling from height; other accident
MeSH Terms: conditions — Wounds and Injuries; Stress Disorders, Post-Traumatic | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Dietary Supplement: Omega-3 Polyunsaturated Fatty Acid
  Interventions: Dietary Supplement: Omega-3 Polyunsaturated Fatty Acid
- 2 (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 Polyunsaturated Fatty Acid — A capsule of omega-3 Polyunsaturated Fatty Acid, 300mg (including 70% docosahexaenoic acid, 7% eicosapentaenoic acid and other), 7 capsules per day in 12 week.
  Arms: 1
Dietary Supplement: Placebo — Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of Polyunsaturated Fatty Acid for the prevention of Posttraumatic Stress Disorder (PTSD) in patients with accidental injuries.

DETAILED DESCRIPTION:
Accidental injuries, mostly motor vehicle accident, in civilian population are frequent events.For instance, nearly one-third of injured patients appear to develop trauma-related psychiatric illness and the major diagnoses are post-traumatic stress disorder (PTSD) and depressive disorder.Omega-3 Polyunsaturated Fatty Acid (Omega-3 PUFA) has some evidence of efficacy of treatment in patients with anxiety and mood disorders, but no evidence of preventing anxiety and mood disorders that occur subsequent to accidental injuries.We evaluate efficacy and safety of Omega-3 PUFA for the secondary prevention of Posttraumatic Stress Disorder (PTSD) and related psychiatric illness in patients with accidental injury

ELIGIBILITY:
Inclusion Criteria:

1. 18 plus years
2. A native Japanese speaking ability
3. Possibility to contact patients with injury in 240 hours, and dosing in oral use
4. Physical and metal status to possible understands scope and contents in the trial and gets informed consent

Exclusion Criteria:

1. Clearly irretrievable acute brain parenchyma damage and subdural or subarachnoidal bleeding detected by computed tomography and/or magnetic resonance imaging
2. Cognitive impairment: Mini Mental State Examination < 24
3. Heavy drinker or 100IU/L ≦ γGTP in administration
4. Heavy smoker (over 40 cigarettes per day)
5. History and current suspicion in diagnosis of psychosis and bipolar I disorder
6. Suspicion in diagnosis of alcoholic, substance-related disorder and eating disorder
7. Existence of marked serious symptoms such as suicidal ideation, self-harm behavior, dissociation, status of need rapidly psychiatric treatment
8. Use of anti-epilepsy drug, lithium, ethyl icosapentate and anti-coagulant drug (for example, aspirin, warfarin, etc) within 3 month at regular intervals
9. Use of polyunsaturated fatty acid supplement within 3 month at regular intervals
10. Habit of eating fish over 4 times per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2008-12; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Total score of Clinician-Administrated PTSD Scale | Three month

SECONDARY OUTCOMES:
Incidence of diagnosis of PTSD (including partial PTSD) | Three month, one month
Total score of Montgomery Asberg Depression Rating Scale (MADRAS) | Three month, one month
Incidence of depression evaluated by Mini-International Neuropsychiatric Interview (MINI) | Three month, one month
Autonomic response measured before, during and after script driven imagery and acoustic stimulation | Three month
Score of Impact of Event Scale revised (IES-R) | Three month, one month
Score of Hospital Anxiety and Depression scale (HADS) | Three month, one month
Score of health related Quality of Life scale, SF-36 | Three month, one month
Score of Conner-Davidson Resilience Scale (CD-RISC) | Three month, one month
Brain-derived neurotrophic factor (BDNF) in serum | Three month, one month
Number of days of leave taken from the time of injury | Three month
Buss-Perry Aggression Questionnaire (BAQ) | Three month, one month, baseline
Total score of Clinician-Administrated PTSD Scale (CAPS) | One month
DHEA: dehydroepiandrosterone | Three month, one month
NPY: neuropeptide Y | Three month, one month
IL-1 beta: interleukin 1 beta | Three month, one month
IL-6: interleukin 6 | Three month, one month
TNF alpha: tumor necrosis factor alpha | Three month, one month
D-serine | Three month, one month
L-serine | Three month, one month
DL-serine | Three month, one month
Activin | Three month, one month

CONTACTS AND LOCATIONS:
Overall Officials: Yutaka Matsuoka, M.D.,Ph.D., Principal Investigator — National Disaster Medical Center, Tachikawa, Tokyo ,Japan
Locations (1):
- National Disaster Medical Center, Tachikawa, Tokyo, Japan

REFERENCES:
- [Background] Matsuoka Y, Nishi D, Yonemoto N, Hamazaki K, Matsumura K, Noguchi H, Hashimoto K, Hamazaki T. Tachikawa project for prevention of posttraumatic stress disorder with polyunsaturated fatty acid (TPOP): study protocol for a randomized controlled trial. BMC Psychiatry. 2013 Jan 5;13:8. doi: 10.1186/1471-244X-13-8. PMID 23289548
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for prevention of post-traumatic stress disorder (PTSD) in individuals experiencing acute traumatic stress symptoms. Cochrane Database Syst Rev. 2024 May 20;5(5):CD013613. doi: 10.1002/14651858.CD013613.pub2. PMID 38767196
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for universal prevention of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2022 Feb 10;2(2):CD013443. doi: 10.1002/14651858.CD013443.pub2. PMID 35141873
- [Derived] Matsuoka Y, Nishi D, Hamazaki K, Yonemoto N, Matsumura K, Noguchi H, Hashimoto K, Hamazaki T. Docosahexaenoic acid for selective prevention of posttraumatic stress disorder among severely injured patients: a randomized, placebo-controlled trial. J Clin Psychiatry. 2015 Aug;76(8):e1015-22. doi: 10.4088/JCP.14m09260. PMID 26335087
- [Derived] Matsuoka Y, Nishi D, Tanima Y, Itakura M, Kojima M, Hamazaki K, Noguchi H, Hamazaki T. Serum pro-BDNF/BDNF as a treatment biomarker for response to docosahexaenoic acid in traumatized people vulnerable to developing psychological distress: a randomized controlled trial. Transl Psychiatry. 2015 Jul 7;5(7):e596. doi: 10.1038/tp.2015.89. PMID 26151924